CLINICAL TRIAL: NCT01719380
Title: A Phase Ib/II Multi-center, Open-label, Dose Escalation Study of LGX818 and Cetuximab or LGX818, BYL719, and Cetuximab in Patients With BRAF Mutant Metastatic Colorectal Cancer
Brief Title: Study of LGX818 and Cetuximab or LGX818, BYL719, and Cetuximab in BRAF Mutant Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818X2103; C4221002 (Other: Alias Study Number); 2012-002138-35 (EudraCT Number)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
Keywords: Open-label dose escalation; BRAF inhibitor; LGX818; PI3K inhibitor; BYL719; EGFR; cetuximab; metastatic colorectal cancer; KRAS; BRAF; V600
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab; Alpelisib

ARMS (2):
- LGX818 + cetuximab (Experimental)
  Interventions: Drug: LGX818; Drug: Cetuximab
- LGX818 + BYL719 + cetuximab (Experimental)
  Interventions: Drug: LGX818; Drug: Cetuximab; Drug: BYL719

INTERVENTIONS:
Drug: LGX818
Drug: Cetuximab
Drug: BYL719
  Arms: LGX818 + BYL719 + cetuximab

SUMMARY:
This study will assess the safety and efficacy of LGX818 when combined with cetuximab or combined with cetuximab and BYL719 in patients with BRAF mutant metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* Progression after at least one prior standard of care regimen or be intolerant to irinotecan-based regimens
* Life expectancy ≥ 3 months
* ECOG performance status ≤ 2

Exclusion Criteria:

* Symptomatic or untreated leptomeningeal disease
* Symptomatic brain metastasis
* Patients with clinically manifested diabetes
* Acute or chronic pancreatitis
* Clinically significant cardiac disease

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-11-23 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- United States (29):
  - Keck Hospital of USC, Los Angeles, California
  - LAC&USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA University of California Los Angeles, Los Angeles, California
  - Westwood Bowyer Clinic, Peter Morton Medical Building, Los Angeles, California
  - UCLA Hematology Oncology, Santa Monica, California
  - UCLA Santa Monica Medical Center & Orthopaedic Hospital, Santa Monica, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at North Haven, North Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - University of Utah - Huntsman Cancer Institute - PPDS, Salt Lake City, Utah
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Redwood Health Center - ARUP Lab Draw Location, Salt Lake City, Utah
  - John A Moran Eye Center, Salt Lake City, Utah
- Royal Melbourne Hospital, Parkville, Victoria, Australia
- UZ Gasthuisberg, Leuven, Vlaams Brabant, Belgium
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- France (2):
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - EDOG - Institut Claudius Regaud - PPDS, Toulouse
- Germany (2):
  - University Hospital of Koln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen
- Ospedaliero Universitaria di Modena Policlinico, Modena, Italy
- Japan (2):
  - Pharmacy of National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Netherlands (3):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Oslo Myeloma Center - PPDS, Oslo, Norway
- South Korea (2):
  - Samsung Medical Center - PPDS, Gangnam-Gu, Seoul Teugbyeolsi
  - Asan Medical Center - PPDS, Songpa-Gu, Seoul Teugbyeolsi
- Spain (3):
  - Instituto de Investigacion Oncologica Vall d'Hebron (VHIO) - EPON, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in two phases Phase 1b and Phase 2. Phase 1b of the study was dose escalation phase to determine maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of LGX818 in combination with cetuximab (dual combination) and of LGX818 in combination with BYL719 and cetuximab (triple combination). Phase 2 of the study was to determine the clinical efficacy and safety of dual and triple combination in study participants.
Groups:
- Phase 1b: LGX818 100 mg + Cetuximab: Participants received 100 mg of LGX818 (encorafenib) orally once daily along with cetuximab orally once weekly in each cycle of 28 days continuously, until disease progression (PD), unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 200 mg + Cetuximab; Phase 2: LGX818 200 mg + Cetuximab: Participants received 200 mg of LGX818 orally once daily along with cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 400 mg + Cetuximab: Participants received 400 mg of LGX818 orally once daily along with cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 450 mg + Cetuximab: Participants received 450 mg of LGX818 orally once daily along with cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab: Participants received 200 mg of LGX818 along with 100 mg of BYL719 (alpelisib) orally once daily and cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab: Participants received 200 mg of LGX818 along with 200 mg of BYL719 orally once daily and cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab; Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab: Participants received 200 mg of LGX818 along with 300 mg of BYL719 orally once daily and cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
- Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab: Participants received 300 mg of LGX818 along with 200 mg of BYL719 orally once daily and cetuximab orally once weekly in each cycle of 28 days continuously, until PD, unacceptable toxicity, withdrawal of informed consent or death, whichever occurred first. Participants were followed up to 30 days after last dose of study treatment (up to a maximum duration of 43 months).
Period: Overall Study
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Started | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 52
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 51
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 4 | 3
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Participant/Guardian Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 2 | 6 | 5 | 6 | 3 | 7 | 10 | 6 | 39 | 42
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab | Total
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 52 | 156
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 1 | 4 | 7 | 5 | 2 | 4 | 8 | 6 | 32 | 38 | 107
  >=65 years | 1 | 3 | 2 | 3 | 1 | 4 | 2 | 1 | 18 | 14 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 6 | 4 | 1 | 5 | 7 | 5 | 36 | 27 | 96
  Male | 0 | 4 | 3 | 4 | 2 | 3 | 3 | 2 | 14 | 25 | 60

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Incidence of Dose Limiting Toxicities (DLTs): Cycle 1
Description: DLTs were defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the first 28 days of treatment and meets any of the criteria included blood and lymphatic system disorders, investigations (blood, renal, hepatic, metabolic), skin and subcutaneous tissue disorders: rash, HFSR (hand foot skin reaction) and/or photosensitivity, metabolism and nutrition disorders: hyperglycemia, gastrointestinal disorders, cardiac disorders, vascular disorders, general disorders and administration site conditions, tumor lysis syndrome, ophthalmologic and other adverse events: study drug-related fever, alkaline phosphatase elevation.
Time Frame: Cycle 1: Day 1 to Day 28
Population: The dose-determining set consisted of all participants from the phase 1b safety set who either met the following minimum exposure criterion and had scheduled safety evaluations or discontinued earlier due to DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 8 | 7 | 3 | 7 | 9 | 7
Participants | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1

2. Primary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause. Participants who did not progress per RECIST (Response Evaluation Criteria in Solid Tumors) version (v) 1.1, were not known to have died prior to the data cut-off, or received any further anticancer therapy were censored at the date of last adequate tumor assessment or the anticancer therapy date, whichever was earlier.
Time Frame: From the date of randomization until the first documentation of disease progression or death due to any cause, censored date, whichever occurred first (maximum up to 43 months)
Population: The full analysis set 2 (FAS2) comprised of all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 50 | 52
months | 4.2 [3.0 to 5.1] | 4.9 [4.0 to 7.1]

3. Secondary Outcome: Number of Participants With Treatment - Emergent Adverse Events of Grade 3 or 4 Severity Based on National Cancer Institute of Common Terminology Criteria (NCI-CTCAE), Version 4.0
Description: An AE was any untoward medical occurrence attributed to study drug in participants who received study drug. As per NCI-CTCAE v4.0, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to study drug. Treatment-emergent AEs are between first dose of study drug and up to 30 days after last dose of study drug, that were absent before treatment or that worsened relative to pretreatment state. Number of participants with any Grade 3 or 4 treatment-emergent AE were reported in this outcome measure.
Time Frame: From screening up to 30 days after the last dose of study treatment (for a maximum duration of 43 months, approximately)
Population: The safety set included all participants from the full analysis set who received at least 1 dose of LGX818 (encorafenib), BYL719 (alpelisib) or cetuximab and had at least 1 valid post baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 52
Participants | 2 | 4 | 6 | 7 | 3 | 5 | 7 | 6 | 33 | 43

4. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of LGX818 (Encorafenib)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: The PK analysis set consisted of all participants who had at least one blood sample providing evaluable PK data, received at least 1 dose of study drug, and experienced no major protocol deviations with relevant impact on the PK data. Here 'Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 6 | 8 | 5 | 3 | 8 | 6 | 4 | 15 | 15
liter per hour | 16.8 (3.60) | 11.7 (6.10) | 12.1 (5.95) | 12.3 (4.96) | 7.69 (3.13) | 14.2 (5.75) | 14.1 (3.65) | 17.8 (17.4) | 13.1 (5.07) | 10.9 (5.70)

5. Secondary Outcome: Apparent Total Plasma Clearance at Steady State (CL/F, ss) of LGX818 (Encorafenib)
Description: Clearance of a drug at steady state is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: The PK analysis set consisted of all participants who had at least one blood sample providing evaluable PK data, received at least 1 dose of study drug, and experienced no major protocol deviations with relevant impact on the PK data. Here 'number analyzed' signifies number of participants evaluable for each specified category and 'Overall Number of Participants Analyzed' signifies number of participants with at least one PK sample analyzed.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 6 | 28 | 36
liter per hour
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 8 | 10 | 4 | 0 | 0
  Cycle 1 Day 8 |  |  |  |  | 17.0 (3.42) | 24.4 (18.3) | 15.4 (4.25) | 22.4 (17.7) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 4 | 4 | 6 | 3 | 6 | 7 | 2 | 10 | 12
  Cycle 2 Day 1 | 13.9 (4.72) | 31.1 (11.9) | 31.6 (2.19) | 30.5 (12.3) | 32.6 (6.88) | 20.2 (7.91) | 22.7 (5.68) | 38.4 (16.4) | 28.2 (8.97) | 23.3 (11.6)

6. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of BYL719 (Alpelisib)
Description: as for outcome 4
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: The PK analysis set consisted of all participants who had at least 1 blood sample providing evaluable PK data, received at least 1 dose of study drug, and experienced no major protocol deviations with relevant impact on the PK data. Here 'Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 5 | 7 | 4 | 10
liter per hour | 12.7 (2.03) | 12.1 (3.96) | 11.6 (1.85) | 11.7 (5.38) | 15.6 (9.61)

7. Secondary Outcome: Apparent Total Plasma Clearance at Steady State (CL/F, ss) of BYL719 (Alpelisib)
Description: as for outcome 5
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: The PK analysis set consisted of all participants who had at least 1 blood sample providing evaluable PK data, received at least 1 dose of study drug, and experienced no major protocol deviations with relevant impact on the PK data. Here 'number analyzed' signifies number of participants evaluable for each specified category and 'Overall Number of Participants Analyzed' signifies number of participants with at least one PK sample analyzed.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 36
liter per hour
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 9 | 2 | 0
  Cycle 1 Day 8 | 16.5 (5.96) | 13.2 (2.29) | 13.7 (7.20) | 11.6 (6.05) |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 2 | 7
  Cycle 2 Day 1 | 18.3 (0.794) | 10.3 (1.23) | 12.5 (1.60) | 19.0 (6.51) | 17.9 (10.5)

8. Secondary Outcome: Apparent Terminal Volume of Distribution (Vz/F) of LGX818 (Encorafenib)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 6 | 8 | 5 | 3 | 8 | 6 | 4 | 15 | 15
liter | 104 (28.3) | 60.3 (25.8) | 62.8 (31.8) | 57.2 (29.6) | 49.2 (12.4) | 75.7 (31.6) | 64.6 (20.6) | 60.7 (44.0) | 63.5 (29.9) | 80.9 (93.9)

9. Secondary Outcome: Apparent Terminal Volume of Distribution at Steady State (Vz/F, ss) of LGX818 (Encorafenib)
Description: Volume of distribution at steady state is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F, ss) is influenced by the fraction absorbed.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 6 | 28 | 36
liter
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 8 | 10 | 4 | 0 | 0
  Cycle 1 Day 8 |  |  |  |  | 78.4 (13.0) | 98.2 (84.5) | 78.6 (26.2) | 88.8 (53.6) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 4 | 4 | 6 | 3 | 6 | 7 | 2 | 10 | 11
  Cycle 2 Day 1 | 66.8 (13.7) | 131 (45.8) | 110 (41.1) | 142 (84.5) | 137 (32.9) | 91.6 (41.4) | 102 (39.9) | 187 (89.5) | 117 (37.6) | 105 (42.2)

10. Secondary Outcome: Apparent Terminal Volume of Distribution (Vz/F) of BYL719 (Alpelisib)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 5 | 7 | 4 | 10
liter | 112 (22.0) | 104 (31.0) | 105 (34.3) | 106 (78.6) | 123 (50.7)

11. Secondary Outcome: Apparent Terminal Volume of Distribution at Steady State (Vz/F, ss) of BYL719 (Alpelisib)
Description: Volume of distribution at steady state was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F, ss) is influenced by the fraction absorbed.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 36
liter
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 9 | 2 | 0
  Cycle 1 Day 8 | 110 (40.7) | 97.0 (20.6) | 105 (30.2) | 82.5 (18.8) |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 2 | 6
  Cycle 2 Day 1 | 138 (20.7) | 75.4 (11.2) | 104 (10.7) | 144 (44.5) | 149 (100)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of LGX818 (Encorafenib)
Description: Tmax was defined as the time to reach maximum observed plasma concentration of encorafenib.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 6 | 9 | 7 | 3 | 8 | 9 | 5 | 17 | 21
hour | 2.00 [1.98 to 2.02] | 1.99 [0.97 to 2.05] | 2.03 [1.00 to 4.00] | 2.17 [1.00 to 5.97] | 1.00 [0.98 to 1.98] | 2.02 [1.00 to 4.02] | 2.00 [0.87 to 5.95] | 3.87 [1.50 to 4.13] | 2.00 [0.93 to 6.12] | 2.03 [0.50 to 8.00]

13. Secondary Outcome: Time to Reach Maximum Plasma Concentration at Steady State (Tmax, ss) of LGX818 (Encorafenib)
Description: Tmax, ss was defined as the time to reach maximum observed plasma concentration of LGX818 (encorafenib) at steady state.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 6 | 28 | 36
hour
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 8 | 10 | 5 | 0 | 0
  Cycle 1 Day 8 |  |  |  |  | 0.98 [0.75 to 4.00] | 1.98 [1.00 to 3.98] | 2.00 [1.12 to 4.02] | 3.92 [0.50 to 4.08] |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 5 | 6 | 7 | 3 | 7 | 8 | 3 | 11 | 14
  Cycle 2 Day 1 | 1.51 [1.00 to 2.02] | 2.00 [1.00 to 4.03] | 1.98 [0.97 to 4.00] | 1.98 [1.05 to 2.05] | 2.00 [1.00 to 2.02] | 2.02 [1.05 to 6.00] | 3.00 [1.92 to 7.98] | 2.27 [2.07 to 3.97] | 1.15 [0.98 to 5.93] | 2.00 [1.88 to 6.00]

14. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of BYL719 (Alpelisib)
Description: Tmax was defined as the time to reach maximum observed plasma concentration of alpelisib.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 8 | 5 | 15
hour | 1.98 [0.98 to 2.00] | 3.97 [1.93 to 6.00] | 2.00 [0.87 to 5.95] | 2.10 [1.50 to 4.50] | 2.05 [1.92 to 8.00]

15. Secondary Outcome: Time to Reach Maximum Plasma Concentration at Steady State (Tmax, ss) of BYL719 (Alpelisib)
Description: Tmax, ss was defined as the time to reach maximum observed plasma concentration of BYL719 (alpelisib) at steady state.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 36
hour
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 8 | 9 | 5 | 0
  Cycle 1 Day 8 | 1.97 [1.00 to 4.00] | 3.99 [1.00 to 7.97] | 2.15 [1.12 to 4.02] | 4.07 [0.00 to 4.10] |
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 7 | 8 | 4 | 9
  Cycle 2 Day 1 | 2.02 [1.00 to 4.00] | 4.00 [1.05 to 6.00] | 3.93 [2.00 to 5.98] | 4.03 [3.97 to 8.00] | 2.02 [1.00 to 6.00]

16. Secondary Outcome: Time of Last Observed Plasma Concentration (T-last) of LGX818 (Encorafenib)
Description: T-last was defined as the time to reach last observed plasma concentration of encorafenib.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 6 | 9 | 7 | 3 | 8 | 9 | 5 | 17 | 21
hour | 23.98 [23.98 to 23.98] | 23.69 [8.00 to 24.00] | 24.03 [22.33 to 24.83] | 23.58 [8.80 to 24.13] | 23.00 [22.52 to 24.30] | 23.06 [7.97 to 24.22] | 22.02 [8.47 to 24.37] | 23.87 [8.23 to 25.92] | 23.85 [8.00 to 24.25] | 23.50 [5.38 to 24.50]

17. Secondary Outcome: Time of Last Observed Plasma Concentration at Steady State (T-last, ss) of LGX818 (Encorafenib)
Description: T-last, ss was defined as the time to reach last observed plasma concentration of encorafenib at steady state.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 6 | 28 | 36
hour
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 8 | 10 | 5 | 0 | 0
  Cycle 1 Day 8 |  |  |  |  | 23.78 [23.75 to 23.92] | 23.36 [7.58 to 23.98] | 23.92 [23.48 to 23.97] | 23.87 [21.83 to 23.95] |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 5 | 6 | 7 | 3 | 7 | 8 | 3 | 11 | 14
  Cycle 2 Day 1 | 23.89 [23.88 to 23.90] | 22.13 [7.30 to 23.85] | 14.05 [6.00 to 24.67] | 23.45 [6.00 to 23.98] | 23.97 [7.25 to 24.20] | 23.08 [8.00 to 23.98] | 23.94 [7.00 to 24.38] | 23.42 [22.08 to 23.58] | 23.80 [8.07 to 24.17] | 23.42 [8.00 to 24.48]

18. Secondary Outcome: Time of Last Observed Plasma Concentration (T-last) of BYL719 (Alpelisib)
Description: T-last was defined as the time to reach last observed plasma concentration of alpelisib.
Time Frame: Cycle 1 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 8 | 5 | 15
hour | 23.00 [22.52 to 24.30] | 23.06 [7.97 to 24.22] | 22.76 [8.47 to 24.37] | 23.87 [8.23 to 25.92] | 23.17 [7.92 to 24.50]

19. Secondary Outcome: Time of Last Observed Plasma Concentration at Steady State (T-last, ss) of BYL719 (Alpelisib)
Description: T-last, ss was defined as the time to reach last observed plasma concentration of alpelisib at steady state.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 8 | 10 | 6 | 36
hour
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 8 | 9 | 5 | 0
  Cycle 1 Day 8 | 23.78 [23.75 to 23.92] | 23.36 [7.58 to 23.98] | 23.87 [7.75 to 23.97] | 23.87 [21.83 to 23.95] |
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 7 | 8 | 4 | 9
  Cycle 2 Day 1 | 23.97 [7.25 to 24.20] | 23.08 [8.00 to 23.98] | 23.94 [7.00 to 24.38] | 23.47 [22.08 to 23.58] | 23.77 [7.00 to 25.50]

20. Secondary Outcome: Plasma Trough Concentration at Steady State (Ctrough, ss) of LGX818 (Encorafenib)
Description: Ctrough, ss was defined as plasma trough concentration of encorafenib at steady state.
Time Frame: Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 5 | 6 | 6 | 3 | 7 | 8 | 1 | 11 | 15
nanogram per milliliter | 9.87 (6.69) | 20.5 (28.0) | 15.7 (22.0) | 20.6 (18.4) | 7.69 (1.76) | 10.4 (5.05) | 26.5 (31.4) | 29.2 (NA) — Standard deviation was not estimated as only 1 participant was analyzed. | 9.24 (5.19) | 15.0 (17.8)

21. Secondary Outcome: Plasma Trough Concentration at Steady State (Ctrough, ss) of BYL719 (Alpelisib)
Description: Ctrough, ss was defined as plasma trough concentration of alpelisib at steady state.
Time Frame: Cycle 2 Day 1: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 +/- 2 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 3 | 7 | 8 | 1 | 8
nanogram per milliliter | 36.7 (21.0) | 108 (41.1) | 283 (156) | 66.0 (NA) — Standard deviation was not estimable as only 1 participant was analyzed. | 141 (76.5)

22. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization or date of start of treatment to the date of death due to any cause or data censoring date, whichever occurred first. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From the date of randomization or date of start of treatment to the date of death due to any cause or data censoring date, whichever occurred first (up to 43 months)
Population: The FAS1 comprised all participants who received at least 1 full or partial dose of their assigned combination of study drugs during Phase 1b. The FAS2 comprised all randomized participants in Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 52
months | 15.0 [14.8 to 15.2] | 5.4 [1.2 to 7.8] | NA [2.9 to NA] — Median and upper limit of 95% Confidence Interval (CI) were not estimable due to fewer participants with event. | 16.6 [3.9 to 23.5] | 6.6 [5.0 to NA] — Upper limit of 95% CI was not reached at the time of data cut-off. | 8.7 [3.8 to 27.1] | 9.8 [3.7 to 25.2] | NA [5.3 to NA] — Median and upper limit of 95% Confidence Interval (CI) were not estimable due to fewer participants with event. | 9.3 [5.8 to 15.6] | 8.5 [6.1 to 15.2]

23. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate as assessed by the investigator per RECIST v1.1, was defined as percentage of participants with a best overall response of complete response (CR) or partial response (PR), were recorded from date of randomization or date of start of treatment until date of first documentation of progressive disease (PD) or death due to any cause. CR was defined as complete disappearance of all target and non-nodal target lesions, and sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Only confirmed CR and PR are counted (those confirmed at least 4 weeks).
Time Frame: From date of randomization or date of start of treatment until date of first documentation of PD or death due to any cause (maximum up to 43 months)
Population: The FAS 1 comprised all participants who received at least 1 full or partial dose of their assigned combination of study drugs during Phase 1b. The FAS2 comprised all randomized participants in Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7 | 50 | 52
percentage of participants | 50.0 [1.3 to 98.7] | 14.3 [0.4 to 57.9] | 11.1 [0.3 to 48.2] | 25.0 [3.2 to 65.1] | 33.3 [0.8 to 90.6] | 25.0 [3.2 to 65.1] | 20.0 [2.5 to 55.6] | 0 [0.0 to 41.0] | 24.0 [13.1 to 38.2] | 26.9 [15.6 to 41.0]

24. Secondary Outcome: Duration of Response (DOR)
Description: DOR: Time between date of the first documented response (CR or PR) and the date of first documented PD or death due to underlying cancer. If PD or death due to underlying cancer not occurred, then participant was censored at the date of last tumor assessment other than unknown. DOR was calculated for responders (confirmed) only. CR: Disappearance of all target, non-target lesions sustained for >=4 weeks and any pathological lymph nodes reduced in short axis to <10mm. PR: >=30% decrease in sum of diameters of target lesions, taking as reference baseline sum of diameter. PD for target lesions: At least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study treatment, with absolute increase of >=5 mm, or appearance of >=1 new lesions. PD for non-target lesions: Unequivocal progression of pre-existing lesions/increase in overall tumor burden leading to discontinuation of therapy or appearance of new unequivocal malignant lesion.
Time Frame: From the first documentation of OR (confirmed CR or PR) to first documentation of PD/death due to any cause or censoring date, whichever occurred first (up to 43 months)
Population: The FAS 1 comprised all participants who received at least 1 full or partial dose of their assigned combination of study drugs during Phase 1b. The FAS2 comprised all randomized participants in Phase 2. Here 'Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 11 | 14
months | 10.6 [NA to NA] — CI values were not estimated due to single participant. | 2.3 [NA to NA] — CI values were not estimated due to single participant. | 21.7 [NA to NA] — CI values were not estimated due to single participant. | 8.1 [5.4 to 10.9] | 3.9 [NA to NA] — CI values were not estimated due to single participant. | 3.6 [2.8 to 4.4] | 3.3 [2.8 to 3.8] |  | 5.6 [2.0 to NA] — Upper limit of 95% CI was not estimable due to low numbers of participant with events. | 5.3 [2.7 to 10.8]

25. Secondary Outcome: Time to Response (TTR)
Description: TTR as assessed by investigator according to RECIST v1.1, was defined as the time (in months) from date of randomization or date of start of treatment until first documented response (CR or PR) or data censoring date, whichever occurred first. CR was defined as complete disappearance of all target and non-target lesions sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants who did not achieve a confirmed PR or CR, were censored at last adequate tumor assessment date when they did not progress (including deaths not due to underlying disease) or at maximum follow-up (from study start to study end date) when participant had an event for progression-free survival.
Time Frame: From the date of randomization or date of start of treatment until first documented response (CR or PR) or data censoring date, whichever occurred first (maximum up to 43 months)
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 12 | 15
months | 2.8 [NA to NA] — CI values were not estimated due to single participant. | 1.4 [NA to NA] — CI values were not estimated due to single participant. | 3.9 [NA to NA] — CI values were not estimated due to single participant. | 4.0 [1.4 to 6.7] | 1.5 [NA to NA] — CI values were not estimated due to single participant. | 3.5 [1.4 to 5.6] | 2.0 [1.4 to 2.5] |  | 1.7 [1.2 to 7.7] | 1.5 [1.4 to 1.7]

26. Secondary Outcome: Phase 1b: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. Participants who did not progress per RECIST v1.1, were not known to have died prior to the data cut-off, or received any further anticancer therapy were censored at the date of last adequate tumor assessment or the anticancer therapy date, whichever was earlier.
Time Frame: From date of start of treatment to the date of event defined as the first documented progression or death due to any cause, censored date, whichever occurred first (maximum up to 43 months)
Population: The FAS 1 comprised all participants who received at least 1 full or partial dose of their assigned combination of study drugs during Phase 1b.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab
Number analyzed (Participants) | 2 | 7 | 9 | 8 | 3 | 8 | 10 | 7
months | 12.0 [10.6 to 13.4] | 3.7 [1.2 to 4.1] | 2.8 [1.3 to 4.3] | 12.0 [1.8 to 12.3] | 5.4 [4.4 to 9.1] | 4.3 [3.8 to 13.6] | 4.1 [1.7 to 5.8] | 4.2 [2.9 to 12.3]

27. Secondary Outcome: Phase 2: Number of Participants With Any Variant in Gene Status at Baseline
Description: Gene alterations/expression relevant to the RAF/MEK/ERK (proto-oncogene serine/threonine-protein kinase/ mitogen-activated ERK kinase/ extracellular signal-regulated kinases) and EGFR/PI3K/AKT (epidermal growth factor receptor/ phosphatidylinositol 3-kinase/ protein kinase B) pathways in tumor tissue, baseline molecular status (mutation/amplification/expression) in tumor tissue of potential predictive markers of tumor response or resistance i.e. BRAF (v-raf murine sarcoma viral oncogene homolog B1), HRAS (harvey rat sarcoma protein), KRAS (V-Ki-ras2 kirsten rat sarcoma viral oncogene homolog B1), NRAS (neuroblastoma RAS viral oncogene homolog), PTEN (phosphatase and tensin homolog), PIK3CA (phosphatidylinositol 3-kinase gene), MAP2K1 (mitogen-activated protein kinase 1), MAP2K2 (mitogen-activated protein kinase 2), ARAF, c-MET, RAF1, EGFR was analyzed.
Time Frame: Baseline (Day 1)
Population: The FAS2 comprised all randomized participants in Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Number analyzed (Participants) | 50 | 52
Participants | 30 | 34

ADVERSE EVENTS:
Time Frame: From screening up to 30 days after the last dose of study treatment (maximum up to 43 months)
Description: Same event may appear as both AE and SAE. An event may be categorized as serious in 1 participant and non-serious in other, or participant may experience both SAE and non-SAE. The safety set included all participants from the FAS who received at least one dose of LGX818 (encorafenib), BYL719 (alpelisib) or cetuximab and had at least one valid post baseline safety assessment.
Arm/Group | Phase 1b: LGX818 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + Cetuximab | Phase 1b: LGX818 400 mg + Cetuximab | Phase 1b: LGX818 450 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab | Phase 2: LGX818 200 mg + Cetuximab | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab
Serious Adverse Events (participants affected / at risk) | 2/2 | 5/7 | 6/9 | 6/8 | 2/3 | 5/8 | 6/10 | 4/7 | 25/50 | 33/52
Other Adverse Events (participants affected / at risk) | 2/2 | 7/7 | 9/9 | 8/8 | 3/3 | 8/8 | 10/10 | 7/7 | 50/50 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: LGX818 100 mg + Cetuximab (N=2) | Phase 1b: LGX818 200 mg + Cetuximab (N=7) | Phase 1b: LGX818 400 mg + Cetuximab (N=9) | Phase 1b: LGX818 450 mg + Cetuximab (N=8) | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab (N=3) | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab (N=8) | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab (N=10) | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab (N=7) | Phase 2: LGX818 200 mg + Cetuximab (N=50) | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab (N=52)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 5 | 5
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 3
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Thrombosis in device (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: LGX818 100 mg + Cetuximab (N=2) | Phase 1b: LGX818 200 mg + Cetuximab (N=7) | Phase 1b: LGX818 400 mg + Cetuximab (N=9) | Phase 1b: LGX818 450 mg + Cetuximab (N=8) | Phase 1b: LGX818 200 mg + BYL719 100 mg + Cetuximab (N=3) | Phase 1b: LGX818 200 mg + BYL719 200 mg + Cetuximab (N=8) | Phase 1b: LGX818 200 mg + BYL719 300 mg + Cetuximab (N=10) | Phase 1b: LGX818 300 mg + BYL719 200 mg + Cetuximab (N=7) | Phase 2: LGX818 200 mg + Cetuximab (N=50) | Phase 2: LGX818 200 mg + BYL719 300 mg + Cetuximab (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 8 | 12
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 4
Eye irritation (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 4 | 0 | 4 | 7 | 3 | 17 | 25
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 0 | 4 | 8 | 5 | 23 | 30
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 4 | 1 | 3 | 1 | 2 | 17 | 21
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 0 | 0 | 2 | 2 | 14 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 4 | 0 | 7 | 5 | 5 | 14 | 29
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 3 | 1 | 5 | 18
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 5 | 5 | 1 | 2 | 6 | 3 | 25 | 27
Chills (General disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 2
Malaise (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 3 | 12 | 11
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 8
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 5 | 5
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 3 | 6
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Haemophilus bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 2 | 0 | 0 | 1 | 0 | 5 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 1 | 3 | 1 | 5 | 3 | 2 | 9 | 19
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 5 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 5 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 5
Blood iron decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 16 | 7
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 6 | 3
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 3
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 4 | 16 | 19
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 2 | 3 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 3 | 2 | 3 | 4 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 6 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 4 | 4 | 5 | 18
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 3 | 1 | 1 | 0 | 1 | 12 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3 | 0 | 2 | 1 | 1 | 8 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 8 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 19 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 4 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 5 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4 | 1 | 6
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 3 | 1 | 0 | 1 | 1 | 2 | 17 | 13
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 6 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 4 | 7
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis in device (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 7 | 8
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 3 | 0 | 1 | 2 | 2 | 8 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 2 | 1 | 8 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 2 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 3 | 1 | 2 | 4 | 2 | 9 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 0 | 4 | 1 | 4 | 9 | 15
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 4 | 2 | 1 | 9 | 12
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 3 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 2 | 11
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 7 | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 5
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 4 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Distichiasis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trichomegaly (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Accommodation disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 4
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Adverse event (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 7
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fear (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bloody discharge (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group performance status improved (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macular reflex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fine motor skill dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.